CLINICAL TRIAL: NCT01079104
Title: Hepa Wash Treatment of Patients With Hepatic Dysfunction in Intensive Care Units
Acronym: HEPATICUS-2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The foundations of our pilotstudy planning has changed.
Sponsor: Hepa Wash GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS002
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Liver Dysfunction; Critical Illness
Keywords: Liver failure; Hepatic insufficiency; Artificial liver; Albumin dialysis
MeSH Terms: conditions — Liver Diseases; Critical Illness; Liver Failure; Hepatic Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Standard Medical Therapy
  Interventions: Procedure: Standard Medical Therapy
- Hepa Wash (Experimental): Treatment with the liver support system "Hepa Wash"
  Interventions: Device: Hepa Wash

INTERVENTIONS:
Device: Hepa Wash — Intervention frequency: 1-10 treatments (decision of the investigator)
  Duration of intervention per patient: Treatment until recovery or death (max. 6 weeks)
  Other Names: Hepa Wash procedure; the HIP1001 system
  Arms: Hepa Wash
Procedure: Standard Medical Therapy — Standard of care treatment
  Arms: Control

SUMMARY:
Patients with hepatic dysfunction are known to have a high mortality rate. Hepa Wash(R) is a newly developed liver and renal support system that is based on the use of recycled albumin dialysate. The new system has shown a high detoxification capacity in in-vitro and preclinical studies. The aim of the study is to evaluate the safety and efficacy of the Hepa Wash system in patients with hepatic dysfunction in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

1. Bilirubin ≥ 2 mg/dl AND
2. SOFA-score ≥ 9 calculated 12 hours after initiating medical resuscitation measures AND
3. Patient is in the intensive care unit AND
4. Signed informed consent of the patient or legal representative AND
5. Patients are 18 years or older AND
6. Enrollment of patients within 96 hours of fulfilling inclusion criteria (1-3).

Exclusion Criteria:

1. Patient with known history of chronic liver disease
2. Untreatable extrahepatic cholestasis
3. Patient has a survival prognosis of less than 6 weeks because of a chronic disease (e.g. metastasizing cancer) and before the acute event which lead to the ICU admission.
4. PaO2/FIO2 ≤ 100 mmHg
5. Patients on kidney dialysis
6. Patients with MELD-score of 40
7. Mean arterial pressure ≤ 50 mmHg despite conventional medical treatment
8. Patient testament excludes the use of life-prolonging measures
9. Post-operative patients whose liver failure is related to liver surgery
10. Uncontrolled seizures
11. Active or uncontrolled bleeding
12. Weight ≥ 120 kg
13. Pregnancy
14. Patient diagnosed with Creutzfeldt-Jakob disease
15. Participation in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-09; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
30-day mortality rate | 30 days
  Mortality 30 days after the first intervention

SECONDARY OUTCOMES:
Multiorgan system failure according to the Sequential Organ Failure Assessment (SOFA) Score | 72 hours
  The Sequential Organ Failure Assessment (SOFA) Score analyses the severity of illness according to 6 organ systems (CNS, Liver, Kidney, Hemodynamic, Coagulation, Lung). Each system is given 0 to 4 points for a total of 24 points. A value >2 in each of the systems indicates organ failure. An overall value > 14 indicates 90% probability of in-hospital mortality.
Adverse Events | 30 days
  Adverse Events during the intervention will be assessed
Number of days on ventilation | 30 days
  Number of days with need of mechanical ventilation after first intervention
Number of days without extracorporeal treatment | 30 days
  Number of days without the need of extracorporeal renal and/or liver replacement therapy after the first intervention
180d-mortality rate | 180 days
  Mortality 180 days after the first intervention
1y-mortality rate | 1 year
  Mortality 1 year after the first intervention

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Huber, PD Dr., Principal Investigator — II Medizinische Klinik, Klinikum rechts der Isar, Munich
Locations (1):
- II Medizinische Klinik, Klinikum rechts der Isar, Munich, Bavaria, Germany

REFERENCES:
- [Result] Huber W, Henschel B, Schmid R, Al-Chalabi A. First clinical experience in 14 patients treated with ADVOS: a study on feasibility, safety and efficacy of a new type of albumin dialysis. BMC Gastroenterol. 2017 Feb 16;17(1):32. doi: 10.1186/s12876-017-0569-x. PMID 28209134